CLINICAL TRIAL: NCT06693414
Title: Effect of Health Promotion Education on Healthy Life Awareness, Salutegenic Health Indicators and Health Literacy
Brief Title: Health Promotion Education, Healthy Life Awareness, Salutogenic Health Indicators and Health Literacy
Acronym: HeProHeLiSIHL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Sultan Ayaz Alkaya, Professor, Gazi University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 24.09.2024/15
Record Dates: First submitted 2024-11-13; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Salutogenesis; Health Literacy; Health Status Measures
Keywords: nursing students; health promotion; nursing intervention; salutogenetic health indicators; general health literacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group: Health promotion education (Experimental): A 14-week health promotion program will be implemented for the intervention group. The training will use lecture, question-and-answer, individual work, and group work techniques. Additionally, activities targeting health-promoting behaviors will be conducted.
  Interventions: Other: Tailored health promotion education; Other: Routine nursing education
- Control group: routine nursing education group (Active Comparator): Participants in the control group will not receive additional health promotion training apart from vocational training.
  Interventions: Other: Routine nursing education

INTERVENTIONS:
Other: Tailored health promotion education — 14 weeks tailored education
  Arms: Intervention group: Health promotion education
Other: Routine nursing education — 14 weeks nursing education

SUMMARY:
Health promotion is a comprehensive process that includes supporting knowledge, skills, and environmental conditions to improve the health levels of individuals and communities. In nursing practice, health promotion plays a critical role in guiding, educating, and raising awareness among individuals about health. Learning foundational knowledge in health promotion allows first-year nursing students to provide more informed and effective health counseling as they gain clinical experience. Enhancing health awareness among first-year nursing students is vital not only for their personal health but also for their future professional competency. Developing awareness of healthy living can positively influence students' health behaviors, empowering them to make more informed health decisions. Awareness of healthy living habits also helps students acquire knowledge in areas such as stress management, nutrition, exercise, and sleep, which can improve their performance in clinical practice. Moreover, nursing students' level of health literacy is crucial for sustaining health behaviors throughout life. Nurses with high health literacy are better equipped to interpret health information effectively, leading to more informed decisions in patient care and healthcare delivery. Therefore, it is essential that nursing students have a high level of health literacy, as it is necessary for their personal development and for maintaining the health of the individuals they serve. Salutogenesis is an approach that focuses on the factors that support and enhance health rather than simply the absence of disease. This approach emphasizes the active role individuals play in maintaining and improving their health. Thus, it is believed that developing salutogenic health perspectives in nursing students from the beginning of their education is important. This study will be conducted to determine the effects of education aimed at health promotion on nursing students' awareness of healthy living, salutogenic health indicators, and health literacy.

DETAILED DESCRIPTION:
Health promotion is a comprehensive process that includes the support of knowledge, skills, and environmental conditions to improve the health levels of individuals and communities. The World Health Organization (WHO) defines health promotion as the process of enabling people to increase control over and improve their health (WHO, 1986). This approach goes beyond disease prevention and embraces a concept of health that includes physical, mental, and social well-being (Nutbeam, 2000). Health promotion helps individuals adopt healthy lifestyles and positively change their health-related behaviors. It also aims to reduce health inequalities and enables communities to establish sustainable health policies (Green & Tones, 2010). In nursing practices, health promotion plays a critical role in guiding individuals, educating them, and raising awareness about health.

Emphasizing the importance of health promotion at the start of nursing education is crucial for the professional development of nursing students. Health promotion not only encourages individuals to adopt healthy lifestyles but is also an important step in preventing and improving diseases (Pender et al., 2015). Learning the fundamentals of health promotion during their first year will enable nursing students to provide more informed and effective health counseling in their future clinical experiences (Edelman & Mandle, 2018). Furthermore, establishing a strong foundation in protecting and promoting individual and community health supports nurses in providing sustainable health services throughout their careers (Whitehead, 2004). Thus, health promotion not only enhances the quality of patient care but also contributes to the mission of protecting public health.

Developing healthy living awareness among first-year nursing students is of great importance for both their individual health and their future professional competencies. Healthy living awareness positively influences students' health behaviors, helping them make more informed health decisions (Whitney, 2018). Awareness of healthy living habits also enables students to gain knowledge about stress management, nutrition, exercise, and sleep, allowing them to perform better in clinical practice (Lenz, 2017). Therefore, developing this awareness at an early stage is essential for individual health sustainability and professional growth. Additionally, acquiring healthy lifestyle habits during their student years allows nurses to guide their future patients more effectively (Pender et al., 2015). In this context, health literacy is highly significant in maintaining health behaviors throughout life.

Health literacy refers to individuals' ability to understand, evaluate, and use health-related information, and developing this skill is critically important for first-year nursing students (Ayaz-Alkaya & Terzi, 2019; Akca & Ayaz-Alkaya, 2021). Nurses with a high level of health literacy can interpret health information more effectively, making more informed decisions in patient care and health service delivery (Nutbeam, 2008). Developing this skill in the early years of nursing education equips students to be more prepared for future clinical practice and to successfully guide patient education (Berkman et al., 2011; Sorensen et al., 2012). Therefore, a high level of health literacy is necessary for nursing students both for their individual development and to sustain the health of those they serve.

Salutogenesis is an approach that considers health not merely as the absence of disease but focuses on factors that support and strengthen an individual's health. This concept, developed by Aaron Antonovsky, seeks to explain how individuals can protect their health by increasing their resilience to stress (Antonovsky, 1979). The salutogenesis model is based on the idea that health is a continuous process and evaluates individuals' capacity to cope with stressors through their abilities to comprehend, manage, and find meaning (Lindström & Eriksson, 2005). In health promotion, this approach is known to empower individuals to take an active role in maintaining and improving their health. Salutogenesis is particularly used as a guide in nursing for care and education models that promote healthy living habits in individuals (Eriksson & Lindström, 2008). It is considered important to foster the salutogenic health of nursing students starting from their school years.

A review of the literature reveals no studies specifically focused on improving salutogenic health and health literacy levels in first-year nursing students. This study aims to draw attention to the importance of the topic.

ELIGIBILITY:
Inclusion Criteria:

* being 18 and older years old
* studying in nursing department
* being voluntary to participate in
* speaking Turkish as a mother language

Exclusion Criteria:

* having any visual and/or hearing disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 232 (Estimated)
Dates: Start 2024-11-20 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Healthy life awareness | 14 weeks up to December
  The Healthy Life Awareness Scale (HeLAS) was developed by Özer and Yılmaz to determine the healthy life awareness level among individuals (Özer & Yılmaz, 2020). It is a 5-point Likert-type scale (1:totally disagree-5:totally agree) with fifteen items and four sub-dimensions. The total score can be got from the scale ranges between 15 and 75. There is no cut-off point; the higher the score, the more awareness of healthy life increases. The Cronbach's alpha of the total scale is 0.81 (Özer & Yılmaz, 2020).
Salutogenetic health indicators | 14 weeks up to December
  The scale developed by Bringsen and colleagues in 2009, and validated and tested for reliability in Turkish by Acı and colleagues (2024), aims to achieve a salutogenic and holistic perspective in measuring health through health indicators. The scale includes questions related to experience, morale, tension, sleep, concentration, creativity, problem-solving, expression of emotions, illness, energy level, social capacity, and physical function. It consists of 12 items on a 6-point Likert scale and has two sub-dimensions: personal characteristics and interactive function. There are no reverse items on the scale. Participants' views over the past 4 weeks are assessed. Scores on the scale range from 12 to 72. The higher the score, the better the individual's health from a salutogenic perspective. In the scale's validity and reliability study, the Cronbach's alpha reliability coefficient was found to be 0.91 (Acı et al., 2024).
Health literacy | 14 weeks up to December
  The HLS19-Q12 is a 12-item short version of the 47-item European Health Literacy Scale, developed by Pelikan and colleagues on behalf of the HLS19 Consortium of the WHO Action Network M-POHL team to assess health literacy levels in the general adult population (Pelikan et al., 2022). The Turkish validity and reliability study of the scale was conducted by Terzi and colleagues (Terzi et al., 2024). The scale is onedimensional and in Likert format, with responses ranging from '1=very difficult, 2=difficult, 3=easy, 4=very easy, 99=don't know.' The total score is calculated as a percentage by dividing the number of questions answered as 'easy' or 'very easy' by the number of valid responses and multiplying by 100. Only responses of '1=very difficult, 2=difficult, 3=easy, 4=very easy' are considered valid and included in score calculation. In the validity and reliability study of the scale, the Cronbach's alpha coefficient was found to be 0.886 (Terzi et al., 2024).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Terzi H, Akca A, Ayaz-Alkaya S. Adaptation of the health literacy survey19-Europe-Q12 into Turkish culture: A psychometric study. J Eval Clin Pract. 2024 Dec;30(8):1782-1790. doi: 10.1111/jep.14161. Epub 2024 Oct 7. PMID 39373230
- [Background] Aci OS, Gencbas D, Ciydem E, Kackin O. Validity and reliability study of the Turkish version of the Salutogenic Health Indicator Scale. Int J Nurs Pract. 2024 Apr;30(2):e13231. doi: 10.1111/ijn.13231. Epub 2023 Dec 20. PMID 38123188